CLINICAL TRIAL: NCT05315557
Title: Efficacy and Safety of Vasopressin Versus Terlipressin as a Second Vasopressor in Critically Ill Cirrhotics With Septic Shock- the VITEL-C Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-48
Record Dates: First submitted 2022-03-07; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Septic Shock; Cirrhosis, Liver
MeSH Terms: conditions — Shock, Septic; Liver Cirrhosis | interventions — Terlipressin; Vasopressins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terlipressin (Experimental): Terlipressin 1mg/24 hours
  Interventions: Drug: Terlipressin
- Vasopressin (Active Comparator): Vasopressin 0.03 U/hour
  Interventions: Drug: vasopressin

INTERVENTIONS:
Drug: Terlipressin — 1mg/24 hour and titrate according to MAP
  Arms: Terlipressin
Drug: vasopressin — 0.03 U/hour and titrate according to MAP
  Arms: Vasopressin

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by dysregulated host response. A Subset of sepsis is septic shock which has almost 4-6 times the mortality when compared to sepsis. Septic shock has underlying cellular and metabolic abnormalities in addition to circulatory dysfunction. The circulatory dysfunction in sepsis is in the form of severe vasodilatation with high cardiac index. Cirrhosis is a state of hyperdynamic circulation. The mortality of septic shock in these group of patients is still higher.

At the onset of septic shock there is initially an increased secretion of Arginine vasopressin. However, this initial rise is short lasting, and the vasopressin levels come back to normal or low serum levels with continued hypotension. However, even normal levels are too low for the degree of hypotension in septic shock. This causes a relative deficiency of vasopressin in septic shock. The exact time when this fall happens is not known and it is likely to be variable. Vasopressin was therefore tried as an agent in septic shock. Terlipressin is a synthetic analogue of vasopressin. It has a greater selectivity for the V1 receptor. Terlipressin is also shown to be effective in septic shock in cirrhotics3. Other vasoactive agents are not preferred in cirrhotics - dopamine due to high risk of arrhythmias and dobutamine as baseline cardiac output of cirrhotics is high which further increases in sepsis and dobutamine would further add to it. However, it may be given in myocardial dysfunction. Noradrenaline is recommended as the first vasopressor to be started in general in septic shock population. No study has compared the effectiveness of vasopressin and Terlipressin when added to noradrenaline in patients with cirrhosis. Acute kidney injury is a very common complication of septic shock in cirrhotics.

DETAILED DESCRIPTION:
Hypothesis: We hypothesise that vasopressin would be non-inferior to terlipressin as a second vasopressor in critically ill cirrhotics with septic shock and would have lesser adverse effects when compared to terlipressin.

Aim: To compare the efficacy of adding continuous infusion of terlipressin versus vasopressin to noradrenaline in causing improvement in systemic hemodynamics and microcirculation.

Methodology:

Study population:

1. Critically ill cirrhotic - Defined as a cirrhotic patient who presents with at least one organ failure, defined by SOFA score WITH
2. septic shock - Defined as a patient in septic shock after initial fluid resuscitation and antibiotic administration, requiring a noradrenaline of at least 2.6mcg/min to maintain a MAP more than 65mmHg.

Study design: Prospective open label randomised controlled study. The study will be conducted in Department of Hepatology ILBS- intensive care unit.

Study period: 1 year

Sample size: Based on the previous studies it is assumed that terlipressin + noradrenaline group would give a response rate of 93%, it was assumed that vasopressin and noradrenaline would give a response rate 15% less than the terlipressin and noradrenaline group and a response rate of 78% was assumed. Further considering an alpha error of 5% and power 95% with a non-inferiority margin of 10% we need to enroll 82 cases Assuming a 10% dropout rate we need to enroll 90 cases with 45 in each arm. However, we decided to enroll 100 cases randomized into 2 groups, 50 each by block randomization method by taking a block size of 10

Patients will be evaluated in the Emergency Room. Detailed history and clinical examination and investigation accordingly will be sent when septic shock is clinically suspected

Fluid Resuscitation Initially a 16G peripheral line will be placed. CVP line and arterial line preferably in the radial artery will be placed as soon as possible.

5% albumin will be used as the resuscitation fluids according to the FRISC protocol.

Fluid response will be assessed at the end of 1 hour

Antibiotics Antibiotics will be given according to the institutional policy

Vasopressors Noradrenaline will be started at a dose of 0.05mcg/kg/min and titrated. All the infusions will be given via central line placed in the jugular, subclavian or femoral vein by a critical care expert under USG guidance.

Intervention:Patients after screening for all exclusion criteria will be randomised into 2 arms (group-1, Terlipressin arm) and (group-2, Vasopressin arm) in a ratio 1:1

* STATISTICAL ANALYSIS: Continuous data- Student's t test
* Nonparametric analysis- Mann Whitney test
* Survival outcome By Kaplan-Meier method curve.
* For all tests, p≤ 0.05 will be considered statistically significant.
* Analysis will be performed using SPSS.
* The analysis will be done with intention to treat and per protocol analysis if applicable.

Stopping rule: Side effects or toxicities that are severe -arrhythmia, AMI, Cardiomyopathy (defined later) Cyanosis.

* Suspicion or confirmed bowel ischemia.
* Patient unwilling for further hospital stay.
* Study unrelated complication here the drug effects could not be assessed (massive
* GI bleed uncontrolled, bowel perforation or any surgical intervention).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70yrs
2. An informed consent from the patient or relative

Exclusion Criteria:

1. Age <18 years and > 70 years
2. Stroke
3. Severe sepsis requiring higher dose of noradrenaline (>1mcg/Kg/min)
4. Myocardial dysfunction, Coronary artery disease, Arrhythmias
5. Peripheral Vascular disease
6. Gut Paralysis
7. Acute on chronic liver failure (ACLF)
8. Hepato-cellular carcinoma (HCC), intrahepatic or extrahepatic malignancy
9. Complete portal vein thrombosis
10. Hepatic vein outflow tract obstruction (HVOTO)
11. Pregnancy
12. Patients with Pa02/FiO2 ratio <150
13. CKD
14. COPD
15. Severe coagulopathy - platelets <20,000 and INR > 4
16. Active Bleed or DIC
17. Patients already on terlipressin or vasopressin in the last 48 hours
18. Extremely moribund patients with an expected life expectancy of less than 24 hours
19. Failure to give informed consent from family members.
20. Patient enrolled in other clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-05 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in systemic hemodynamics at 6 hours after randomization | 6 hours after randomization
  Improvement in systemic hemodynamics defined as discontinuation of noradrenaline infusion OR reversal of shock

SECONDARY OUTCOMES:
Reduction in dose of noradrenaline at the end of 6 hours | 6 hours
Amount of noradrenaline requirements between in each arm at the end of 6 hours | 6 hours
Improvement in Systemic Vascular Resistance (SVR) by 10% or above 500 at 6 hours | 6 hours
  Systemic Vascular Resistance will be measured by using pulmonary thermodilution
Improvement in SVR by 10% or above 500 at 12 hours | 12 hours
Improvement in SVR by 10% or above 500 at 48 hours | 48 hours
Decrease in Cardiac output by 10% or less than 6L after 6 hours of randomization | 6 hour of randomization
  Cardiac output will be measured by using pulmonary thermodilution
KDIGO criteria - increase in urine output in 6 hours | 6 hour
KDIGO criteria - increase in urine output in 12 hours. | 12 hour
KDIGO criteria - increase in urine output in 24 hours | 24 hour
KDIGO criteria - increase in urine output in 48 hours. | 48 hour
improvement in serum creatinine in 24 (Improvement in KDIGO stage at 24) | 24 hour
Improvement in serum creatinine in 48 hours (Improvement in KDIGO stage at 48 hours) | 48 hour
Need of Renal Replacement Therapy | Day 28
Improvement in microcirculation as measured by improvement in lactate | 6 hours
Improvement in microcirculation as measured by improvement in capillary refill time at 6 hours | 6 hours
Improvement in microcirculation as measured by Near IR spectroscopy ina subset of patients whenever feasible | 6 hours
Improvement in microcirculation as measured by improvement in lactate | 24 hours
Improvement in microcirculation as measured by improvement in capillary refill time at 24 hours. | 24 hours
Improvement in microcirculation as measured by Near IR spectroscopy ina subset of patients whenever feasible | 24 hours
Improvement in microcirculation as measured by improvement in lactate | 48 hours
Improvement in microcirculation as measured by improvement in capillary refill time at 48 hours. | 48 hours
Improvement in microcirculation as measured by Near IR spectroscopy ina subset of patients whenever feasible | 48 hours
Improvement in renal resistive index at 24 hours | 24 hours
Improvement in renal resistive index at 48 hours | 48 hours
Incidence of adverse effects till 48 hours after randomization including incidence of rebound hypertension | 48 hours
Mortality at day 28 | Day 28
Days of mechanical ventilation | Day 28
Days of Intensive Care Unit stay. | Day 28
Endothelial function will be measured in a subset of patients | 48 hours
  Endothelial function will be assessed from a change in endothelin-1 and von Willebrand Factor (vWF) levels in a subset of patients whereever feasible
Coagulation function will measure in a subset of patients | 48 hours
  Coagulation function will be measured by change in rotational thromboelastometry test

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided